CLINICAL TRIAL: NCT04556162
Title: Evaluation of Salt Status in Patients With Cystic Fibrosis and the Influence on Nutritional Status and Pulmonary Function. Looking for the Best Surrogate Urinary Markers for Fractional Sodium or Chloride Excretion
Brief Title: Evaluation of Salt Status in Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-05673
Record Dates: First submitted 2020-08-19; First posted 2020-09-21 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Salt; Deficit (or Low); Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fractional sodium excretion — fractional sodium excretion will be compared to urinary sodium/creatinin, sodium/potassium ratio's and sodium concentration.
Other: risk subgroups — subgroup analysis will be performed to identify the patient groups at risk for sodium depletion

SUMMARY:
The results of the annual check-up will be collected to evaluate the best urinary marker for fractional sodium excretion and salt status will be correlated to clinical outcome measures.

DETAILED DESCRIPTION:
Patients with cystic fibrosis need extra salt as they have increased losses through sweat. Current advices are to follow and supplement if needed, however the way to follow salt depletion is unclear.

The best way is to calculate fractional salt excretion. This needs a simultaneous blood and urine sample for electrolytes and creatinin. Urinary surrogate markers have been validated on only 10 patients.

At the annual check-up patients with cystic fibrosis receive these measurements. The investigators will collect the measurements and calculate fractional excretion and the possible surrogate markers on urine. Further this will be correlated to nutritional and pulmonary status and patient subgroups at risk will be identified.

ELIGIBILITY:
Inclusion Criteria:

* all cystic fibrosis patients followed at the Gent University Cystic fibrosis centre
* Providing a paired urine and blood sample at the time of their annual check-up

Exclusion Criteria:

* transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cystic fibrosis patients for whom a complete analysis of both blood and urine is available at the time of their annual check-up
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
fractional sodium excretion (percent) | 1 year
  = (serum creatinin X urinary Sodium)/(plasma sodiumX urinary creatinin)
Urinary sodium/urinary creatinin (mmol/mmol) | 1 year
  calculated based on urinary results
Fractional Chloride excretion (percent) | 1 year
  = (serum creatinin X urinary Chloride)/(plasma Chloride X urinary creatinin)
Fractional Potassium excretion (%) | 1 year
  = (serum creatinin X urinary Potassium)/(plasma PotassiumX urinary creatinin)
ratio urinary sodium/urinary potassium | 1 year
  = calculation of ration urinary sodium/potassium

SECONDARY OUTCOMES:
Body mass index | 1 year
  = Weight/Height X Height expressed as SD of the local population based on Flemish growth charts
Forced expiratory volume in 1 second | 1 year
  measured with lungfunction testing expressed as % of normal for height

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Van Biervliet, MD, PhD, Principal Investigator — Gent University hospital
Locations (1):
- Gent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No